CLINICAL TRIAL: NCT03126955
Title: Microvascular Decompression for HELPS Syndrome: What is the Best Diagnostic Test?
Brief Title: Diagnostic Test of Choice for HELPS Syndrome
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Christopher Honey, Professor & Neurosurgeon, University of British Columbia
Other Study IDs: H17-00953
Record Dates: First submitted 2017-04-10; First posted 2017-04-25 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: HELPS Syndrome
Keywords: microvascular decompression, Xth nerve

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HELPS Syndrome unable to lateralize contractions: Each patient will have the following 3 diagnostic pre-operative tests: i) MRI (CISS sequence), ii) video laryngoscopy, and iii) sequential Botox injections in their throat (left side and then 3 months later on the right side).
  Interventions: Diagnostic Test: Pre-Operative CISS-MRI Sequences; Diagnostic Test: Pre-Operative Interictal Laryngoscopy; Diagnostic Test: Pre-Operative Unilateral and Contralateral Botox

INTERVENTIONS:
Diagnostic Test: Pre-Operative CISS-MRI Sequences — Compare pre-operative MRI diagnosis to intra-operative findings on if both are in agreement
Diagnostic Test: Pre-Operative Interictal Laryngoscopy — Compare pre-operative laryngoscopy diagnosis to intra-operative findings on if both are in agreement
Diagnostic Test: Pre-Operative Unilateral and Contralateral Botox — Compare pre-operative diagnosis using Botox to intra-operative findings on if both are in agreement
  Other Names: Injections spaced 3-months apart

SUMMARY:
Our team recently described a new medical condition called HELPS (Hemi-Laryngo-Pharyngeal-Spasm) syndrome(1). HELPS syndrome is a condition caused by a blood vessel pinching the nerve rootlets of the Vagus nerve (Xth cranial nerve). It is similar to the well recognized hemifacial spasm syndrome but the nerve involved is the Vagus instead of the Facial nerve. As a result, the symptoms are episodic throat contractions and cough. The throat contractions become stronger and more frequent over the years and can lead to a terrifying inability to breath. Patients may end up intubated in the Emergency Department or with a tracheostomy because of inability to breath during a severe episode. Some but not all of our patients can tell which side of their throat (left or right) contracts during a choking episode. In between these choking episodes, patients feel normal. A surgical cure for these patients is Microvascular Decompression of the Xth nerve.

DETAILED DESCRIPTION:
The treatment of HELPS syndrome begins with the correct diagnosis. Some patients are able to localize the side of their symptoms in HELPS syndrome while others are unable to. The purpose of this study is to prospectively study which of the following is the diagnostic test of choice for patients who are unable to localize their HELPS: 1. CISS MRI sequences, 2. interictal laryngoscopy, and 3. unilateral and contralateral Botox injections separated 3-months apart.

Both neuroradiologist and otolaryngologist will be blinded to the outcome of surgery and be asked "based on your diagnostic test, which side do you believe we should perform MVD surgery?"

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with HELPS as described in our initial publication (Honey et al. 2016)
* Patients unable to localize the side of their HELPS syndrome

Exclusion Criteria:

- Unable to provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HELPS (Hemi-Laryngo-Pharyngeal Spasm) Syndrome
  -Subgroup of patients who are unable to localize lateralization of throat contractions
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2017-04-30 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Pre-Operative CISS MRI (One month before surgery) compared to Intraoperative Findings | Pre-Operative and Intra-Operative
  Determine if CISS MRI sequence lateralization in concordance with intraoperative findings
Pre-Operative Interictal Laryngoscopy (One month before surgery) compared to Intraoperative Findings | Pre-Operative vs. Intra-Operative
  Determine if interictal laryngoscopy in concordance with intraoperative findings
Pre-Operative 3 and 6-month Botox Injections compared to Intraoperative Findings | Pre-operative 3 and 6 months vs. Intra-Operative
  Determine if unilateral vs contralateral Botox-induced symptom reduction in concordance with intraoperative findings

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R Honey, MD, DPhil, FRCSC, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Honey CR, Gooderham P, Morrison M, Ivanishvili Z. Episodic hemilaryngopharyngeal spasm (HELPS) syndrome: case report of a surgically treatable novel neuropathy. J Neurosurg. 2017 May;126(5):1653-1656. doi: 10.3171/2016.5.JNS16308. Epub 2016 Jul 8. PMID 27392269